CLINICAL TRIAL: NCT00282100
Title: A Pilot Study of Adjuvant Therapy of Gefitinib (Iressa, ZD1839) in Patients With Resectable Hepatocellular Carcinoma
Brief Title: Adjuvant Therapy of Gefitinib (Iressa, ZD1839) in Patients With Resectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singapore Cancer Syndicate. (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JS0414; NCT00228501 (obsolete NCT alias)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gefitinib (Iressa) (Experimental): Open label single arm study of Gefitinib (Iressa) 250mg daily as adjuvant therapy in patients with resectable Hepatocellular Carcinoma
  Interventions: Drug: Gefetinib (Iressa)

INTERVENTIONS:
Drug: Gefetinib (Iressa)

SUMMARY:
This research is being done to find how soon the liver cancer may come back and whether proteins or genes in tumor, blood or urine can give us clues of early recurrence.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common cancers in the world1. HCC risk increases drastically in patients with chronic hepatitis B infection, hepatitis C infection or liver cirrhosis. HCC is very prevalent in our region due to endemic hepatitis B infection and increasing incidence of hepatitis C.

Patients with HCC have very poor prognosis because HCC tumors are usually non-symptomatic. Most patients will not be diagnosed until the disease has reached an advanced stage. Chemotherapy may offer palliative benefit to some patients with advanced HCC but has not been shown to prolong survival in these patients. HCC patients are in need for innovative and targeted therapies. Therefore, we propose to study gefitinib as an adjuvant therapy in patients with resected HCC.

Gefitinib blocks the function of epidermal growth factor receptor which is a key factor in stimulating liver cancer growth. In mice, gefitinib has been shown to reduce the size of liver cancer. It also had anti tumor activity in patients with various cancers including HCC. Gefitinib can relieve disease-related symptoms in these patients. Overall, gefitinib is a very well tolerated treatment and is suitable for long-term use.

At the time of diagnosis and surgical evaluation, patients with resectable hepatocellular carcinoma will be asked to participate in this study.Patients will be registered after consent form is obtained. Patient is asked to donate tumor tissues, urine and blood samples.Tumor and normal specimens are collected at the time of surgery. After patient recovers from surgery (4-6 weeks) and fulfills the eligibility, patient will receive gefitinib 250 mg p.o. daily for 6 months.

Patient will remain on study till completion of treatment. The following are conditions when your study doctor will remove you from the study or stop the therapy:

1. Interruption of treatment for 4 consecutive weeks due to side effects, which do not resolve.
2. withdraw of consent by patient. ii. Your disease becomes worse. iii. New information that gefitinib treatment is harmful to patients has become available.

Patient will be evaluated at one month, 3 months and 6 months on gefitinib. After that, evaluate patient at least every 3 months for first 2 years, then every 6 months for next 3 years, then yearly afterwards. Draw blood and store sera and urine at the same interval until relapse and/or death. Conduct correlative studies of urine, serum and tumor tissue with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

Pathologically newly diagnosis HCC, which is deemed resectable and resected.

Patient has to start gefitinib within 6 weeks of hepatic resection with full recovery.

Patients with positive resection margin or minimal residual disease (<0.5 cm) are also eligible.

ECOG performance status (PS) 0, 1 or 2

Patient must recover fully from hepatic resection ANC > 1,500/uL SGOT < 5 x UNL (upper normal limits) Plt > 75,000/uL Bilirubin < 2 x UNL Serum albumin ≥ 2.5g/dL

Creatinine < 1.5 mg/dl or 125 u/L, alpha fetoprotein < 50 ug/L

Signed informed consent

Age > 18

No space occupying lesion on CT scan of the liver i.e. normal CT scan post-resection. Small lesion in the liver after resection can be ablated by alcohol injection or radio frequency ablation and can make patient eligible.

Negative pregnancy test of the blood within 7 days of starting treatment in female patient of childbearing potential.

No prior systemic therapy or I131 or chemoembolization treatment after surgery.

Can take or swallow medication orally i.e. no chronic or persistent nausea and vomiting

No other malignancy except for adequately treated basal cell or squamous cell skin cancer or cervical cancer in-situ.

No active infection, symptomatic CHF, unstable angina, uncontrolled cardiac arrhythmia and psychiatric disorder.

No concomitant medications such as phenytoin, carbamazepine, rifampicin, barbiturates, ketoconazole and itraconazole, which are potent inducers of CYP3A4 or potent inhibitors of CYP3A4.

Patient is not taking St. John's Wort.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-12 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
To study the changes of selected genetic or protein markers through the treatment and find out whether some of them can be potential biomarkers for disease relapse. | Minimum 2 years

SECONDARY OUTCOMES:
To evaluate the effect of gefitinib as an adjuvant therapy on recurrence free survival in patients with resectable hepatocellular carcinoma; to evaluate the treatment toxities of genifitib. | Minimum 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, M.D., Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore